CLINICAL TRIAL: NCT04995042
Title: An Open-Label, Multicenter, Dose Escalation And Expansion Study Of SHR7280 In Subjects With Hormone Sensitive Prostate Cancer
Brief Title: A Phase 1 Dose Escalation and Expansion Study Of SHR7280 In Subjects With Hormone Sensitive Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR7280-104
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Hormone Sensitive Prostate Cancer

STUDY DESIGN:
Intervention Model Description: Open-label, Multicenter, Singel Group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR7280 Does Escalation and Expansion (Experimental)
  Interventions: Drug: SHR7280

INTERVENTIONS:
Drug: SHR7280 — Drug: SHR7280 All participants receive SHR7280 alone.

SUMMARY:
This is an open-label, multicenter, dose escalation and expansion Phase 1 study of SHR7280 in adult patients with hormone sensitive prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent document；
2. Age ≥18 years old;
3. Histologically or cytologically confirmed prostate adenocarcinoma;
4. Candidate for androgen deprivation therapy (ADT) for the management of hormone-sensitive prostate cancer；
5. Appropriate serum testosterone and serum PSA concentration at screening as specified in the protocol；
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1;
7. Adequate organ performance based on laboratory blood tests;
8. Agree to use adequate contraception prior to study entry and for the duration of study participation.

Exclusion Criteria:

1. Previously received gonadotropin-releasing hormone analogues (GnRH-a) for more than 12 months total duration (if GnRH-a was received for 12 months or less, then that GnRH-a must have been completed washout period prior to the first dose of study drug).
2. Patients who have received chemotherapy for prostate cancer;
3. History of surgical castration;
4. Received Abiraterone acetate with 3 months prior to the first dose of study drug;
5. Receieved molecular target therapy, immunotherapy, androgen receptor blockade, 5-alpha reductase inhibitors, estrogen, and other investigational compound with 4 weeks prior to the first dose of study drug;
6. Patients with known or suspected brain metastasis；
7. Diagnosis or treatment for another systemic malignancy within 5 years before study treatment initiation;
8. Patients with uncontrolled and clinically significant hypertension and diabetes;
9. Known hypersensitivity to SHR7280, SHR7280 excipients,；
10. History of immunodeficiency (including HIV infection) or organ transplantation;
11. Known active hepatitis B or C infection;
12. Other serious accompanying illnesses, which, in the researcher's opinion, could seriously adversely affect the safety of the treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Adverse Events（AEs） | 30 days after last dose
Dose Limited Toxicity (DLT) | 28 Days (first cycle)
Maximum tolerable dose (MTD) | 28 Days (first cycle）
Recommended dose for phase II (RP2D) | Up to 12 months

SECONDARY OUTCOMES:
Area under the plasma concentration time curve in the dosing interval AUC(TAU) of SHR7280 | 30 days after last dose
Maximum observed plasma concentration (Cmax) of SHR7280 | 30 days after last dose
Observed trough plasma concentration (Ctrough) of SHR7280 | 30 days after last dose
Time of maximum observed plasma concentration (Tmax) of SHR7280 | 30 days after last dose
Serum testosterone concentrations | 30 days after last dose
Serum luteinizing hormone (LH) concentrations | 30 days after last dose
Serum follicle stimulating hormone (FSH) concentrations | 30 days after last dose
Time to Achieve Testosterone Concentrations < 50 ng/dL | 30 days after last dose
Percentage of Participants With Effective Castration Rate Over 24 Weeks | Day 1 of Week 5 to Day 1 of Week 25
Percentage of Participants With Effective Castration Rate Over 48 Weeks | Day 1 of Week 5 to Day 1 of Week 49
Percentage of Serum Prostate-Specific Antigen Concentration Change frome Baseline at the End of Weeks 4, 8, 12 | Day 1 of Weeks 5, 9 and 13
Time to Prostate-Specific Antigen Progression | 30 days after last dose

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided